CLINICAL TRIAL: NCT04717999
Title: Pilot Study of UWNKG2D CAR-T in Treating Patients With Recurrent Glioblastoma
Brief Title: Pilot Study of NKG2D CAR-T in Treating Patients With Recurrent Glioblastoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: UWELL Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UBP-P02-3001-GBM
Record Dates: First submitted 2021-01-16; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UWN2D CAR-T (Experimental)
  Interventions: Biological: NKG2D CAR-T

INTERVENTIONS:
Biological: NKG2D CAR-T — The NKG2D CAR-T will be administrated via intracerebroventricular injection through an Ommaya catheter. Standard treatments such as temozolomide will be stopped during the infusion of NKG2D CAR-T.
  Other Names: UWN2D

SUMMARY:
This is a pilot phase I study to evaluate the safety and efficacy of NKG2D CAR-T cell therapy in patients with relapsed and/or refractory glioblastoma

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed glioblastoma multiforme (GBM) and are at first or second relapse.
* Hemoglobin ≥ 9.0 g/dl, absolute neutrophil count (ANC) ≥ 1,000 cells/µl, platelets ≥ 125,000 cells/µl
* No active infection of HIV, HTLV and Syphilis
* Adequate renal function
* Adequate hepatic function
* Adequate cardiac function
* Adequate venous access for apheresis, and no other contraindications for leukapheresis
* Voluntary informed consent is given.

Exclusion Criteria:

* Pregnant or lactating women.
* Uncontrolled active infection.
* History of hepatitis B or hepatitis C infection.
* Previously treatment with any gene therapy products or cell therapy product in past 28 days.
* Cannot undergo MRI with contrast or SPECT/CT
* HIV infection.
* Have autoimmune disorders
* Have active infection or inflammatory disorders
* Prescreening test results in expansion rate less than 5 folds
* An allergy to gentamycin and/or streptomycin

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who experience a Dose-Limiting Toxicity (DLT) | 2 years
  Defined as the dose safely administered Intratumoral for the treatment of patients with GBM

SECONDARY OUTCOMES:
Overall Response Rate | 1 year
  Defined as the proportion of subjects with overall response of either complete response (CR) or partial response (PR)
Progression-free survival | 1 year
  Defined as date of the first NKG2D CAR-T infusion to the date of disease progression per RANO Response Criteria or death